CLINICAL TRIAL: NCT02949622
Title: Development and Validation of a Multimodal Intervention Program for Patients With Metabolic Syndrome
Brief Title: Multimodal Intervention Program for Patients With Metabolic Syndrome
Acronym: PROMETS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: University Hospital Virgen de las Nieves (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Jaqueline Garcia da Silva, Ph.D. Student, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAPES 5566-10-0
Record Dates: First submitted 2016-10-14; First posted 2016-10-31 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Metabolic Syndrome X
Keywords: Metabolic syndrome; Mediterranean diet; Stress; quality of life; psychological factors
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multimodal intervention program (Experimental): The intervention program will be in group format, with a size of 10 to 12 patients per group and with an extension of 12 sessions. The treatment program will feature sessions with psychoeducation of metabolic syndrome and treatment model, problem solving, stress management, anger management, social skills, self-efficacy and social support.
  Interventions: Behavioral: Multimodal intervention program
- Lifestyle counseling (Active Comparator): The group of lifestyle counseling will have basic guidelines, according to the recommendations of public health.
  Interventions: Other: Lifestyle counseling

INTERVENTIONS:
Behavioral: Multimodal intervention program — The intervention is structured as follows:
  Review of previous session (20 min) Agenda and goals (5 min) Presentation of the topic to be worked (15 min) Training (60 min) Summary and feedback (15 min)
  Arms: Multimodal intervention program
Other: Lifestyle counseling — The group of lifestyle counseling will have basic guidelines, according to the recommendations of public health.
  Arms: Lifestyle counseling

SUMMARY:
The aim of this study is to identify the psychological, emotional and lifestyle variables that can have an influence on the different components of metabolic syndrome (MetS) and develop a program for change lifestyle in this patients.

ELIGIBILITY:
Inclusion Criteria:

* Between 25 and 65 years age
* Waist circumference >88 cm for women and >102 cm for men
* Blood pressure: systolic ≥ 130 mmHg and diastolic ≥ 85 mmHg
* Fasting glucose level ≥ 110mg/dL
* Triglycerides: ≥ 150 mg/dL
* HDL cholesterol ≤40 mg/dL in men and ≤50 mg/DL in women

Exclusion Criteria:

* Osteoarthritis,
* Active inflammatory diseases,
* Severe psychiatric disorders and/or significant cognitive impairment assessed using the Mini-Mental State Examination.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2013-02; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Weight | 2 minutes
  weight (Kg)
Waist circumference | 2 minutes
  (cm). Measured using a tape measure placed in a horizontal plane, located at the midpoint between the last rib and the iliac crest
Blood pressure | 15 minutes
  Taken according to the recommendations of the American Heart Association, and considering the mean of three readings, each separated by two minutes.
Lipid profile | 3 minutes
  lipid profile (HDL-C, total cholesterol, triglycerides)
Glycemic profile (fasting glucose) | 3 minutes
  glycemic profile (fasting glucose)

SECONDARY OUTCOMES:
State-Trait Anger Expression Inventory-2 - STAXI-2 | 5 minutes
  To determine diverse components of anger, such as experience, expression and control, as well as its facets such as state and trait, the Inventory of Expression of Anger State-Trait (STAXI-2) was used. It consists of 49 items organised in 6 scales and 5 subscales, permitting the attainment of an index for each scale and subscale, as well as a general index of the inventory.
Perceived Stress Scale -PSS | 5 minutes
  To measure the perceived stress during the previous month, the Perceived Stress Scale was used, with a total of 14 items.
Assertiveness Inventory | 5 minutes
  To evaluate the general assertiveness, the Assertiveness Inventory (AI) consisting of 30 items was used .
Medical Outcomes Study 12-Item Short Form - SF-12 | 5 minutes
  To determine the health-related quality of life the Medical Outcomes Study 12-Item Short Form (SF-12), which is composed of two components related to physical and mental health, was used.
Mediterranean-diet scale | 5 minutes
  To evaluate the level of adherence to the Mediterranean diet (MedDiet). Consisting of 14 items that evaluate whether foods are included that can prevent cardiovascular risk such as olive oil, fish, vegetables, fruits, cereals and also foods that can increase the chances of risk such as cold meats, trans fats and excess salt. The degree of adherence to the MedDiet is given by the sum of the items. A score below 11 is considered low adherence and higher than 11 as high.
Fagerström Test for Nicotine Dependence | 5 minutes
  To evaluate the degree of physical dependence on nicotine. The test consists of six items with two or four response alternatives. The score ranges from 0 to 10. High scores in the FTND (6 or more) indicate a high degree of dependence.

OTHER OUTCOMES:
Mini Mental State Examination - MMSE | 5 minutes
  To assess the initial mental state of the patient and possible cognitive deficits.
Mini International Neuropsychiatric Interview - MINI | 30 minutes
  Brief diagnostic interview, compatible with the DSM-V and ICD-10 criteria was used to evaluate possible co-morbidities in the sample.
Height | 2 minutes
  height (cm)

CONTACTS AND LOCATIONS:
Locations (1):
- Jaqueline Garcia da Silva, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia-Silva J, Borrego IRS, Navarrete NN, Peralta-Ramirez MI, Aguila FJ, Caballo VE. Efficacy of cognitive-behavioural therapy for lifestyle modification in metabolic syndrome: a randomised controlled trial with a 18-months follow-up. Psychol Health. 2024 Jan-Feb;39(2):195-215. doi: 10.1080/08870446.2022.2055023. Epub 2022 Mar 28. PMID 35345950